CLINICAL TRIAL: NCT02738840
Title: A Post-Market Study Evaluating the Prodigy MRI and Proclaim Elite MR Conditional SCS Systems
Acronym: SCS MRI PMCF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRD_800
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Results first posted 2021-05-24 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: International, multicenter, prospective, and single-arm design
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prodigy MRI or Proclaim Elite MR (Experimental): The Prodigy MRI system is only MR conditional for scans of the head and extremities (upper except shoulder, lower except hip).
  The Proclaim Elite system is MR conditional for scans of the head, extremities or any other body part.
  Interventions: Procedure: MRI scan

INTERVENTIONS:
Procedure: MRI scan — MRI scan

SUMMARY:
A post market study evaluating the safety of the Prodigy MRI and Proclaim Elite MR conditional Spinal Cord Stimulator (SCS) systems.

DETAILED DESCRIPTION:
The study will be performed as an international, multicenter, prospective and single-arm design. The study will be conducted as a Post Market Clinical Follow Up (PMCF) study and the results will be submitted to the Notified Body: BSI Group (BSI).

ELIGIBILITY:
Inclusion Criteria:

* Patient has been implanted with a Prodigy MRI or Proclaim Elite MR conditional SCS system
* Patient will receive an MRI scan in compliance with the Instructions For Use (IFU) for the implanted MR conditional SCS system
* Patient is ≥ 18 years of age
* Patient must be willing and able to comply with study requirements
* Patient must indicate his/her understanding of the study and willingness to participate by signing an appropriate Informed Consent Form

Exclusion Criteria:

* Patient has another implanted device (active or passive) that prohibits safe scanning
* Patient has previously experienced an MRI scan-related adverse event
* Patient is currently enrolled in another Abbott study that collects MRI safety data
* Patient is incapacitated, is unable to read or write, or is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Harbert, Study Director — Abbott
Locations (10):
- United States (3):
  - Napa Valley Orthopedic Medical Group, Napa, California
  - Unity Spine Center, Rochester, New York
  - Clinical Trials of South Carolina, Charleston, South Carolina
- Wilhelminenspital Wien, Vienna, Austria
- AZ Sint-Augustinus, Wilrijk, Belgium
- Germany (2):
  - Medizinische Einrichtungen der Universität Düsseldorf, Dusseldorf, Düsseldorf
  - Hospital Gera -Zentrum für interdisziplinäre Schmerztherapie, Gera, Gera
- Azienda Ospedaliero Universitaria Pisana, Pisa, Italy
- Hospital Virgen de Rocio, Seville, Spain
- Seacroft Hospital, Leeds, Ykshre, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 56 subjects were enrolled at 10 investigational sites in Europe and the United States (US). The first subject was enrolled on 21 October 2016 and the last subject on 22 September 2020. Completion of follow-up occurred on 02 December 2020.
Groups:
- Prodigy MRI or Proclaim Elite MR: The Prodigy MRI system is only MR conditional for scans of the head and extremities (upper except shoulder, lower except hip).
  The Proclaim Elite system is MR conditional for scans of the head, extremities or any other body part.
  MRI scan: MRI scan
Period: Overall Study
Arm/Group | Prodigy MRI or Proclaim Elite MR
Started | 56
Completed | 48
Not Completed | 8
Not completed — MRI Scan not Performed | 5
Not completed — Lost to Follow-up | 1
Not completed — Subject Participation Terminated by Investigator | 1
Not completed — Subject Did not Meet Screening Inclusion/Exclusion Criteria | 1

BASELINE CHARACTERISTICS:
Population: Of the 56 enrolled subjects, 55 subjects completed the baseline visit; one subject did not have an MR conditional Spinal Cord Stimulator (SCS) system implanted.
Arm/Group | Prodigy MRI or Proclaim Elite MR
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Of the 56 enrolled subjects, 55 subjects completed the baseline visit; one subject did not have an MR conditional SCS system implanted.
  years
    number analyzed (Participants) | 55
    (all) | 58.4 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Of the 56 enrolled subjects, 55 subjects completed the baseline visit; one subject did not have an MR conditional SCS system implanted.
  Participants
    number analyzed (Participants) | 55
    Female | 36
    Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 1
  Belgium | 6
  United States | 23
  Italy | 8
  United Kingdom | 5
  Germany | 7
  Spain | 6
IPG type [Count of Participants; unit: Participants] — Population: Of the 56 enrolled subjects, 55 subjects completed the baseline visit; one subject did not have an MR conditional SCS system implanted.
  Participants
    Prodigy MRI: number analyzed (Participants) | 55
    Prodigy MRI | 26
    Proclaim: number analyzed (Participants) | 55
    Proclaim | 29

OUTCOME MEASURES:

1. Primary Outcome: The Rate of the MRI Scan-related Adverse Events
Description: The rate of the MRI scan-related adverse events will be assessed at 1-month follow-up.
Time Frame: 1 month post MRI scan
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: participants
Arm/Group | Prodigy MRI or Proclaim Elite MR
Number analyzed (Participants) | 50
participants | 0

2. Secondary Outcome: Rate of Successful MRI Mode 'Turn on' Functionality
Description: The rate of successful MRI mode 'turn on' functionality will be assessed during pre-MRI scan.
Time Frame: Immediately before MRI Scan
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prodigy MRI or Proclaim Elite MR
Number analyzed (Participants) | 51
percentage of participants
  MRI Mode successfully turned on | 98.0 [89.55 to 99.95]
  MRI Mode not successfully turned on | 2.0 [0.05 to 10.45]

3. Secondary Outcome: Rate of Successful MRI Mode 'Turn Off' Functionality
Description: The rate of successful MRI mode 'turn off' functionality will be assessed during Post-MRI Scan.
Time Frame: Immediately after MRI Scan
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prodigy MRI or Proclaim Elite MR
Number analyzed (Participants) | 50
percentage of participants | 100 [92.89 to 100.00]

4. Secondary Outcome: Rate of Successful 'Turn Off' Functionality for the Stimulation
Description: The rate of successful 'turn off' functionality for the stimulation will be assessed immediately before MRI Scan.
Time Frame: Immediately before MRI Scan
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prodigy MRI or Proclaim Elite MR
Number analyzed (Participants) | 29
percentage of participants | 100 [88.06 to 100.00]

5. Secondary Outcome: Rate of Successful 'Turn on' Functionality for the Stimulation
Description: The rate of successful 'turn on' functionality for the stimulation will be assessed immediately after MRI Scan.
Time Frame: Immediately after MRI Scan
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prodigy MRI or Proclaim Elite MR
Number analyzed (Participants) | 50
percentage of participants | 100 [92.89 to 100.00]

6. Secondary Outcome: Rate of Successful 'Turn on/Off' Functionality for the Stimulation
Description: The rate of successful 'turn on/off' functionality for the stimulation at 1-month follow-up will be assessed.
Time Frame: At 1 month follow-up
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prodigy MRI or Proclaim Elite MR
Number analyzed (Participants) | 27
percentage of participants
  Stimulation successfully turned off | 100 [87.23 to 100.00]
  Stimulation successfully turned on | 100 [87.23 to 100.00]

7. Secondary Outcome: Rate of Successful Adjustments to the Program
Description: The rate of successful adjustments to the program will be assessed. This includes adjustments to stimulation amplitude and switch between stimulation programs.
Time Frame: Immediately before MRI Scan
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prodigy MRI or Proclaim Elite MR
Number analyzed (Participants) | 29
percentage of participants
  Successful adjustments to stimulation amplitude | 100 [88.06 to 100.00]
  Successful switch between stimulation programs: number analyzed (Participants) | 27
  Successful switch between stimulation programs | 100 [87.23 to 100.00]

8. Secondary Outcome: Rate of Successful Adjustments to the Program
Description: as for outcome 7
Time Frame: Immediately after MRI Scan
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prodigy MRI or Proclaim Elite MR
Number analyzed (Participants) | 29
percentage of participants
  Successful adjustments to stimulation amplitude: number analyzed (Participants) | 28
  Successful adjustments to stimulation amplitude | 100 [87.66 to 100.00]
  Successful switch between stimulation programs: number analyzed (Participants) | 24
  Successful switch between stimulation programs | 100 [85.75 to 100.00]

9. Secondary Outcome: Rate of Successful Adjustments to the Program
Description: as for outcome 7
Time Frame: At 1-month follow-up
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prodigy MRI or Proclaim Elite MR
Number analyzed (Participants) | 29
percentage of participants
  Successful adjustments to stimulation amplitude: number analyzed (Participants) | 27
  Successful adjustments to stimulation amplitude | 100 [87.23 to 100.00]
  Successful switch between stimulation programs: number analyzed (Participants) | 27
  Successful switch between stimulation programs | 100 [87.23 to 100.00]

10. Secondary Outcome: Rate of Successful Interrogations and Uploads/Downloads of the Implantable Generators (IPG) Parameters
Description: The rate of interrogations and uploads/downloads of the IPG parameters will be assessed immediately before MRI Scan. This includes establishing a link with the IPG or patient programmer and uploading and downloading of the subject's current program.
Time Frame: Immediately before MRI Scan
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prodigy MRI or Proclaim Elite MR
Number analyzed (Participants) | 29
percentage of participants
  Link successfully established with IPG or Patient Programmer | 100 [88.06 to 100.00]
  Successful upload of subject's current program | 100 [88.06 to 100.00]
  Successful download of subject's current program | 100 [88.06 to 100.00]

11. Secondary Outcome: Rate of Successful Interrogations and Uploads/Downloads of theImplantable Generators (IPG) Parameters
Description: The rate of interrogations and uploads/downloads of the IPG parameters will be assessed immediately after MRI Scan. This includes establishing a link with the IPG or patient programmer and uploading and downloading of the subject's current program
Time Frame: Immediately after MRI Scan
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prodigy MRI or Proclaim Elite MR
Number analyzed (Participants) | 28
percentage of participants
  Link successfully established with IPG or Patient Programmer | 100 [87.66 to 100.00]
  Successful upload of subject's current program | 100 [87.66 to 100.00]
  Successful download of subject's current program | 100 [87.66 to 100.00]

12. Secondary Outcome: Rate of Successful Interrogations and Uploads/Downloads of theImplantable Generators (IPG) Parameters
Description: The rate of interrogations and uploads/downloads of the IPG parameters will be assessed at 1-month follow-up. This includes establishing a link with the IPG or patient programmer and uploading and downloading of the subject's current program
Time Frame: At 1-month follow-up
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prodigy MRI or Proclaim Elite MR
Number analyzed (Participants) | 29
percentage of participants
  Link successfully established with IPG or Patient Programmer: number analyzed (Participants) | 27
  Link successfully established with IPG or Patient Programmer | 100 [87.23 to 100.00]
  Successful upload of subject's current program: number analyzed (Participants) | 25
  Successful upload of subject's current program | 100 [86.28 to 100.00]
  Successful download of subject's current program: number analyzed (Participants) | 25
  Successful download of subject's current program | 100 [86.28 to 100.00]

ADVERSE EVENTS:
Time Frame: 1 month
Description: No serious adverse events or procedure/device-related adverse events were reported in this study.
Arm/Group | Prodigy MRI or Proclaim Elite MR
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT02738840/Prot_SAP_000.pdf